CLINICAL TRIAL: NCT01484210
Title: Phase III Therapeutic Evaluation Study Comparing the Efficacy and Safety of the Fluticasone/Salmeterol (500/50 μg) Combination Administered With Elpenhaler® (Rolenium®) Versus the Innovative One (Seretide Diskus®) in Patients With Asthma.
Brief Title: Single Dose Study of the Fluticasone/Salmeterol (500/50 μg) Administered With Elpenhaler® Versus Diskus®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-FLUSAL-EL-02; 2007-006670-29 (EudraCT Number); Sponsor ID (Other: FLUSAL-02); Sponsor FLUSAL-02 (Other Grant/Funding Number: Elpen Pharmaceutical Co Inc)
Record Dates: First submitted 2011-10-12; First posted 2011-12-02 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2011-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elpenhaler Active - Diskus Placebo (Experimental): Patients on treatment with both devices, Elpenhaler and Diskus, first active substance, second placebo.
  Interventions: Drug: Elpenhaler active - Diskus placebo

INTERVENTIONS:
Drug: Elpenhaler active - Diskus placebo — randomized, double-blind, double-dummy, 2-way crossover, single dose study, comparing the efficacy and safety of the Fluticasone/Salmeterol (500/50 μg) combination administered with Elpenhaler® (Rolenium®) versus the innovative one (Seretide Diskus®) in patients with asthma.

SUMMARY:
The aim of this study is to establish the therapeutic equivalence between the test (Fluticasone/Salmeterol administered with Elpenhaler®, Rolenium®) and the reference formulation (Seretide®, administered with Diskus®), both containing 500/50μg of the Fluticasone/Salmeterol combination.

The study will be conducted in a randomized, double-blind, double-dummy, 2x2 crossover fashion.

DETAILED DESCRIPTION:
In case of inhaled products, it is not possible to follow the classic scheme, based on similarity of plasma concentration-time behavior of parent drug in assessing bioequivalence.

For this reason, a pharmacodynamic study was designed in order to assess the therapeutic equivalence of the new formulation of Fluticasone/Salmeterol with the innovative one. The test and reference Fluticasone/Salmeterol formulations will be compared in terms of their bronchodilator effects in lung function. Forced Expiratory Volume in 1 second (FEV1) will be the primary efficacy measure and will be measured in such a way that a similar time-dependent increase in pulmonary function can be demonstrated for both Fluticasone/Salmeterol formulations in patients with asthma. In terms of safety comparison, repeated measurements of adverse events, vital signs, heart rate, blood hematology and biochemistry as well as ECG changes will enable the establishment of the similar safety profile of the test and reference Fluticasone/Salmeterol combinations.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years,
* diagnosis of asthma of 6 months,
* FEV1 ≥ 50% and ≤ 80% predicted,
* reversibility of at least 12%,
* stable asthma for at least 4 weeks,
* inhaled steroids (ICS) at a stable dose within the previous 30 days,
* PIF 30 - 90 lt/min and
* informed consent.

Exclusion Criteria:

* history of other pulmonary disease,
* asthma exacerbation or respiratory infection within the previous 4 weeks,
* hospitalization for acute asthmatic symptoms requiring parenteral steroids or oral steroid dose increase, within the previous 30 days,
* heavy smokers,
* change of asthma medication within the previous 4 weeks,
* seasonal asthma alone,
* history of severe heart disease,
* pregnancy or lactation,
* use of a β-blocker, of a NSAID or an antiallergic/antihistaminic medication within 2 weeks prior to screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary variable will be the 12-hour average FEV1 [area under the FEV1 versus time curve divided by 12 (FEV1 AUC0-12/12)]. | 0 (baseline), Visit 1 (3-7 days), Visit 2 (3-7 days), Telephone Contact Follow up (3-7 days)
  To establish the therapeutic equivalence between the Fluticasone/Salmeterol combination administered with Elpenhaler® (Rolenium®) and the innovative one (Seretide Diskus®) in terms of their bronchodilator effect in lung function.

SECONDARY OUTCOMES:
The FEV1 values over time for the 12-hour observation period | 0 (baseline), Visit 1 (3-7 days), Visit 2 (3-7 days), Telephone Contact Follow up (3-7 days)
  To compare the efficacy and safety profile of the two Fluticasone/Salmeterol formulations in patients with asthma.
Time to peak FEV1 | 0 (baseline), Visit 1 (3-7 days), Visit 2 (3-7 days), Telephone Contact Follow up (3-7 days)
  To compare the effiacy and safety profile of the two Fluticasone/Salmeterol formulations in patients with asthma
Time to peak FEV1 maximum value | same as FEV1
  same as FEV1

CONTACTS AND LOCATIONS:
Overall Officials: A Dindos, MD, Principal Investigator — Pneumology Surgery, Kojeticka 1021, 27711 Neratovicae
Locations (5):
- Czechia (5):
  - Pneumology surgery Vitezna 201/31, Karlovy Vary, Drahovice
  - Pneumology surgery Vojtesska 237, Kutná Hora, Zizkov
  - Pneumology and allergology surgery Voldusska 750, New Town
  - Pneumology surgery Hostinskeho 1536, Prague
  - Pneumology surgery Generala Janouska 902/17, Prague